CLINICAL TRIAL: NCT06022055
Title: Multimodal Study of the Human Brain Epilepsy Tissue
Acronym: TIPI²
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ICM Co. Ltd. (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP230479
Record Dates: First submitted 2023-05-22; First posted 2023-09-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Focal Drug-resistant Epilepsy
Keywords: Focal drug-resistant epilepsy; Surgery; Biorepository; Biomarkers
MeSH Terms: interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- epileptic patients (Experimental): All patients will be enrolled in the same arm. Patients can be enrolled during the pre-surgical evaluation (group 1) or in the days preceding the surgery (group 2).
  Interventions: Other: Blood and tissue collection

INTERVENTIONS:
Other: Blood and tissue collection — Blood will be collected for group 1 during (i) the enrolment visit, (ii) in the 24 hours following a seizure, (iii)before the surgery and (iv) in the 36 months following the surgery. The left-over tissue, not useful for diagnostic purpose, will be kept for research.
  Blood will be collected for group 2 right before the surgery and in the 36 months following the surgery. The left-over tissue not useful for diagnostic purpose will be kept for research.

SUMMARY:
The TIPI2 study is a blood and tissue collection protocol to create an annotated biorepository to support research in drug-resistant epilepsy.

The aim of the study will be to identify new pathophysiological pathways. For this purpose, the investigators will investigate with a multimodal approach blood and brain samples from patients undergoing a surgery for focal drug-resistant epilepsy. The adult patients will be enrolled either during the pre-surgical evaluation or right before the surgery.

DETAILED DESCRIPTION:
This study aims to investigate blood and brain samples from patients with drug-resistant epilepsy in order to identify new pathophysiological biomarkers.

The investigators will first conduct multimodal research, including:

* electrophysiological analyses
* immunohistochemistry and genetic studies
* biochemistry analyses

Samples will be stored at -80°C for future research.

Patients will undergo a follow-up evaluation within the 36 months following the surgery. New clinical data and biological samples will be collected then.

ELIGIBILITY:
Inclusion Criteria:

* 18 yo or above
* patients with a focal drug-resistant epilepsy
* patients hospitalized for a pre-surgical evaluation or for an epilepsy surgery
* consent obtained from the patient, or legally authorized representative
* affiliated to a social security system

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2037-02-28 (Estimated)

PRIMARY OUTCOMES:
Identification of new pathophysiological mechanisms leading to focal drug-resistant epilepsy : analysis by immuno-histological methods | At the day of surgery; analyses are based on the post-operative tissues
  The investigator will identify inflammatory cells (astrocytes, microglia, lymphocytes and neutrophil polynuclear cells) in the post-operative brain tissue, and will calculate if there is an increase of a part of these cells in the area, defined as the seizure onset zone, as compared to the non-epileptic areas.
Identification of new pathophysiological mechanisms leading to focal drug-resistant epilepsy : analysis by electrophysiological methods | At the day of surgery; analyses are based on the post-operative tissues
  The investigator will record local field potentials and neuronal firing rate from post-operative tissues, and we will research an increase of the rate of interictal epileptiform discharges and of the frequency of the neuronal firing in the seizure-onset zone, as compared to those in non-epileptic areas.
Identification of new pathophysiological mechanisms leading to focal drug-resistant epilepsy : analysis by RNA sequencing methods | At the day of surgery; analyses are based on the post-operative tissues
  The investigator will measure the expression of mRNA in cells of different parts of the post-operative brain tissue, and we will research specific expression of mRNA in the Seizure onset zone, as compared to that in other non-epileptic areas.

SECONDARY OUTCOMES:
Identification of new pathophysiological mechanisms associated with the occurrence of a seizure : analysis of biomarkers by ELISA methods | from inclusion day to 36 months after the surgery
  The investigator will measure several proteins by Elisa, and we will define if there is a specific increase of some proteins in the sample after a seizure, as compared to the level of these proteins far from a seizure.
Identification of new pathophysiological mechanisms associated with an active epilepsy : analysis of biomarkers by ELISA methods | from inclusion day to 36 months after the surgery
  The investigator will measure the different blood cells by flow cytometry, and we will define if there is a specific increase of some cell populations in the sample from epileptic patients, as compared to the level of these cell populations in non-epileptic patients.
Identification of new pathophysiological mechanisms associated with an active epilepsy : analysis of blood cell subtypes by flow cytometry | from inclusion day to 36 months after the surgery
  The investigator will measure the different blood cells by flow cytometry, and we will define if there is a specific increase of some cell populations in the sample from epileptic patients, as compared to the level of these cell populations in non-epileptic patients.
Identification of new pathophysiological mechanisms associated with an active epilepsy : analysis of inflammation biomarkers by digital ultra-sensitive quantitation of proteins methods | from inclusion day to 36 months after the surgery
  The investigator will measure several inflammatory proteins including cytokines, and we will define if there is a specific increase of some proteins in the sample from epileptic patients, as compared to the level of these proteins in non-epileptic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent M. Navarro, MD, PHD, Principal Investigator — APHP
Locations (1):
- Department of Neurology, Epilepsy Unit, Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request
  The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.